CLINICAL TRIAL: NCT00773175
Title: Subcutaneous Rehydration With Hylenex Compared to Intravenous Rehydration in Infants and Young Children With Mild to Moderate Dehydration
Brief Title: Subcutaneous Rehydration Compared to Intravenous Rehydration
Acronym: PEDs-II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HZ2-08-03
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Results first posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-10

CONDITIONS: Dehydration
Keywords: pediatric; hylenex; subcutaneous infusion; hyaluronidase; rHuPH20; recombinant human hyaluronidase
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subcutaneous (Active Comparator): Isotonic fluid rehydration by SC administration with hylenex (150 Units in 1 mL)
  Interventions: Drug: recombinant human hyaluronidase
- Intravenous (Active Comparator): Isotonic fluid rehydration by IV
  Interventions: Drug: recombinant human hyaluronidase

INTERVENTIONS:
Drug: recombinant human hyaluronidase — 150 Units in 1 mL
  Other Names: Hylenex

SUMMARY:
Randomized (1:1 ratio) study of subcutaneous (SC) versus intravenous (IV) fluid rehydration in mildly to moderately dehydrated pediatric patients.

DETAILED DESCRIPTION:
This is a prospective, randomized (1:1 ratio), open-label, parallel group, multicenter, multi-national, study of SC versus IV fluid rehydration in mildly to moderately dehydrated pediatric patients treated in the Emergency Department (ED), inpatient pediatric unit, and/or outpatient urgent care facility. It is expected that up to 186 patients, in order to achieve 148 evaluable patients, will be randomized in a 1:1 ratio to receive isotonic fluid rehydration by either SC administration with hylenex (150 Units) or IV without hylenex.

ELIGIBILITY:
Inclusion Criteria:

* Children of either gender from one month to ≤10 years of age.
* Patients with mild or moderate dehydration
* Healthy child except for the underlying etiology for dehydration
* Pre-dehydration body weight ≥ 5th percentile for age
* Parents or legal guardian(s) available to provide informed consent.

Exclusion Criteria:

* Severe dehydration
* Shock or life-threatening situation (life expectancy < 10 days).
* Requirement for IV access for any indication other than for treatment of dehydration.
* Indwelling IV catheter, except for one intended only for collection of clinical laboratory specimens.
* Any condition precluding SC infusion or infusion site evaluation
* Any reason (prior to study enrollment) for a hospital admission or an extended stay in the ED for other than dehydration.
* Known hypersensitivity to hyaluronidase or hylenex.
* Known hyponatremia (< 130 milliequivalents per liter [mEq/L]) or hypernatremia (> 155 mEq/L).
* Known hypokalemia (< 3.0 mEq/L).
* Any medical condition likely to interfere with the patient's ability to fully complete all protocol-specified interventions, the ability to undergo all protocol-specified assessments, or likely to prolong the patient's need for medical attention beyond that required for treatment of dehydration.
* Participation in an investigational drug or device study within 30 days prior to enrollment in this study.

Ages: 30 Days to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2008-10; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Coburn H Allen, MD, Principal Investigator — Baylor College of Medicine
Locations (25):
- United States (25):
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Tampa General Hospital Children's Medical Center, Tampa, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Children's Healthcare of Atlanta - Scottish Rite, Atlanta, Georgia
  - North Georgia Clinical Research, Dalton, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - Memorial Hospital, South Bend, Indiana
  - University of Louisville, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - William Beaumont Hospital, Troy, Michigan
  - The Children's Mercy Hospital & Clinics, Kansas City, Missouri
  - UMDNJ/Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - St. Joseph's Children's Hospital, Paterson, New Jersey
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - New York Methodist Hospital, Brooklyn, New York
  - Staten Island University Hospital Emergency Department, Staten Island, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Rainbow Children's and Babies Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Dell Children's Medical Center, Austin, Texas
  - Children's Medical Center Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Derived] Spandorfer PR, Mace SE, Okada PJ, Simon HK, Allen CH, Spiro DM, Friend K, Harb G, Lebel F; Increased Flow Utilizing Subcutaneously-Enabled Pediatric Rehydration II (INFUSE-Peds II) Study Group. A randomized clinical trial of recombinant human hyaluronidase-facilitated subcutaneous versus intravenous rehydration in mild to moderately dehydrated children in the emergency department. Clin Ther. 2012 Nov;34(11):2232-45. doi: 10.1016/j.clinthera.2012.09.011. Epub 2012 Oct 11. PMID 23062548

RESULTS

PARTICIPANT FLOW:
Groups:
- Subcutaneous Hylenex: Participants received isotonic fluid rehydration by subcutaneous administration with recombinant human hyaluronidase (hylenex: 150 Units in 1 milliliter [mL]).
- Intravenous Isotonic Fluid: Participants received isotonic fluid rehydration by intravenous injection.
Period: Overall Study
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid
Started | 73 | 75
Initial Fluids Via Randomized Route | 73 | 59
Initial Fluids Via Subcutaneous Rescue (Subcutaneous fluid administration by hylenex-facilitated infusion was given as rescue.) | 0 | 15
No Fluids Received | 0 | 1
Completed | 71 | 73
Not Completed | 2 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Consent Withdrawn | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid | Total
Number analyzed (Participants) | 73 | 75 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.1 (1.72) | 2.4 (2.07) | 2.3 (1.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 36 | 75
  Male | 34 | 39 | 73
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Black or African American | 25 | 22 | 47
  White | 39 | 40 | 79
  Native Hawaiian or Pacific Islander | 0 | 1 | 1
  Unknown | 9 | 12 | 21

OUTCOME MEASURES:

1. Primary Outcome: Mean Total Volume of Fluid Administered at a Single Infusion Site, From the Start to the Cessation of Fluid Administration, for All Randomized Participants
Description: It was anticipated that most participants in this study would be hydrated through only one infusion site. For participants who received fluid at more than one administration site, a single infusion site was defined as the anatomical site at which the majority of the total infusion volume was infused. The term "anatomical site" was designated as: 1) the back; 2) left thigh; 3) right thigh; 4) abdomen; or 5) chest.
Time Frame: During the infusion (single bolus dose of hylenex [1 hr], followed by subcutaneous fluid for 1 hour to 72 hours)
Population: Intent-to-Treat (ITT) Population: all randomly assigned participants for whom the treatment was attempted, (i.e., infusion device placement was initiated)
Measure: Mean (Standard Deviation); unit: milliliters
Groups:
- Subcutaneous Hylenex: Participants received isotonic fluid rehydration by subcutaneous (SC) administration with recombinant human hyaluronidase (hylenex: 150 Units in 1 milliliter [mL]).
- Intravenous Isotonic Fluid: Participants received isotonic fluid rehydration by intravenous (IV) injection.
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid
Number analyzed (Participants) | 73 | 75
milliliters
  Emergency department plus hospital stay | 365.0 (324.57) | 455.8 (597.43)
  Emergency department stay only | 334.3 (226.4) | 299.6 (252.33)
Statistical Analysis 1: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid; Test type: Non-Inferiority — Subcutaneous administration would not be deemed as inferior if the volume infused subcutaneous is ≥85% of the volume infused intravenously; p = 0.5064, ANOVA — P-value for the test of the null hypothesis that the volume delivered via a hylenex-facilitated subcutaneous infusion was ≤85% of the volume delivered intravenously; Emergency department plus hospital stay; Mean Difference (Final Values) = -67.5, 95% CI 2-sided [-221.2 to 86.2] — Treatment difference: subcutaneous minus intravenous
Statistical Analysis 2: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0325, ANOVA — [p-value comment as in outcome 1, analysis 1]; Emergency department stay only; Mean Difference (Final Values) = 24.0, 95% CI 2-sided [-54.6 to 102.7] — Treatment difference: subcutaneous minus intravenous

2. Primary Outcome: Mean Total Volume of Fluid Administered at a Single Infusion Site, From the Start to the Cessation of Fluid Administration, for Non-rescued Participants
Description: It was anticipated that most participants in this study would be hydrated through only one infusion site. For participants who received fluid at more than one administration site, a single infusion site was defined as the anatomical site at which the majority of the total infusion volume was infused. The term "anatomical site" was designated as: 1) the back; 2) left thigh; 3) right thigh; 4) abdomen; or 5) chest. Participants randomized to receive intravenous isotonic fluid were permitted to receive subcutaneous fluid administration by hylenex-facilitated infusion as rescue.
Time Frame: During the infusion (single bolus dose of hylenex [1 hr], followed by subcutaneous fluid for 1 hour to 72 hours)
Population: ITT Population. Only those participants for which fluid administration was initiated were analyzed. Only those participants who did not receive subcutaneous fluid administration by hylenex-facilitated infusion as rescue were analyzed.
Measure: Mean (Standard Deviation); unit: milliliters
Groups:
- Intravenous Isotonic Fluid: Non-rescued: Participants randomized to receive IV isotonic fluid who were not rescued via the hylenex-facilitated SC-rescue route, as IV access could be established.
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid: Non-rescued
Number analyzed (Participants) | 73 | 59
milliliters
  Emergency department plus hospital stay | 365.0 (324.57) | 579.4 (618.49)
  Emergency department stay only | 334.3 (226.4) | 380.8 (223.08)
Statistical Analysis 1: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid: Non-rescued; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.8915, ANOVA — [p-value comment as in outcome 1, analysis 1]; Emergency department plus hospital stay; Mean Difference (Final Values) = -174.7, 95% CI 2-sided [-340.3 to -9.1] — Treatment difference: subcutaneous minus intravenous
Statistical Analysis 2: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid: Non-rescued; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.5469, ANOVA — [p-value comment as in outcome 1, analysis 1]; Emergency department stay only; Mean Difference (Final Values) = -58.6, 95% CI 2-sided [-137.5 to 20.3] — Treatment difference: subcutaneous minus intravenous

3. Primary Outcome: Mean Total Volume of Fluid Administered at a Single Infusion Site, From the Start to the Cessation of Fluid Administration, for All Rescued Participants
Description: as for outcome 2
Time Frame: During the infusion (single bolus dose of hylenex [1 hr], followed by subcutaneous fluid for 1 hour to 72 hours)
Population: ITT Population. Only those participants for which fluid administration was initiated were analyzed. Only those participants randomized to receive intravenous isotonic fluid who received subcutaneous fluid administration by hylenex-facilitated infusion as rescue were analyzed.
Measure: Mean (Standard Deviation); unit: milliliters
Groups:
- Intravenous Isotonic Fluid: SC Rescued: Participants randomized to receive IV isotonic fluid were rescued via the hylenex-facilitated SC-rescue route after IV access could not be established.
Arm/Group | Intravenous Isotonic Fluid: SC Rescued
Number analyzed (Participants) | 15
milliliters
  Emergency department plus hospital stay | 388.3 (281.13)
  Emergency department stay only | 315.3 (150.38)

4. Secondary Outcome: Mean Total Volume of Fluid Administered at All Infusion Sites, From the Start to the Cessation of Fluid Administration, for All Randomized Participants
Description: as for outcome 1
Time Frame: During the infusion (single bolus dose of hylenex [1 hr], followed by subcutaneous fluid for 1 hour to 72 hours)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid
Number analyzed (Participants) | 73 | 75
milliliters
  Emergency department plus hospital stay | 365.4 (324.21) | 455.8 (597.43)
  Emergency department stay only | 334.7 (225.94) | 299.6 (252.33)
Statistical Analysis 1: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.5035, ANOVA — [p-value comment as in outcome 1, analysis 1]; Emergency department plus hospital stay; Mean Difference (Final Values) = -67.0, 95% CI 2-sided [-220.6 to 86.7] — Treatment difference: subcutaneous minus intravenous
Statistical Analysis 2: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0314, ANOVA — [p-value comment as in outcome 1, analysis 1]; Emergency department stay only; Mean Difference (Final Values) = 24.6, 95% CI 2-sided [-54.0 to 103.2] — Treatment difference: subcutaneous minus intravenous

5. Secondary Outcome: Mean Total Volume of Fluid Administered at All Infusion Sites, From the Start to the Cessation of Fluid Administration, for All Randomized Participants Achieving > 200 mL
Description: It was anticipated that most participants in this study would be hydrated through only one infusion site. For participants who received fluid at more than one administration site, a single infusion site was defined as the anatomical site at which the majority of the total infusion volume was infused. The term "anatomical site" was designated as: 1) the back; 2) left thigh; 3) right thigh; 4) abdomen; or 5) chest. The label for hylenex indicated precautionary wording recommending an upper limit on the volume of fluid (200 mL) administered subcutaneously to infants less than 3 years of age. In October 2008, the Food and Drug Administration (FDA) removed this wording from the label, thus negating the need for these data and associated analyses. The protocol was amended to reflect this label change; thus, this analysis was not conducted.
Time Frame: During the infusion (single bolus dose of hylenex [1 hr], followed by subcutaneous fluid for 1 hour to 72 hours)
Population: Randomized Population: all participants who were assigned a patient randomization number
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Mean Total Volume of Fluid Administered at All Infusion Sites, From the Start to the Cessation of Fluid Administration, for Non-rescued Participants Achieving > 200 mL
Description: It was anticipated that most participants in this study would be hydrated through only one infusion site. For participants who received fluid at more than one administration site, a single infusion site was defined as the anatomical site at which the majority of the total infusion volume was infused. The term "anatomical site" was designated as: 1) the back; 2) left thigh; 3) right thigh; 4) abdomen; or 5) chest. Participants randomized to receive intravenous isotonic fluid were permitted to receive subcutaneous fluid administration by hylenex-facilitated infusion as rescue. The label for hylenex indicated precautionary wording recommending an upper limit on the volume of fluid (200 mL) administered subcutaneously to infants less than 3 years of age. In October 2008, the FDA removed this wording from the label, thus negating the need for these data and associated analyses. The protocol was amended to reflect this label change; thus, this analysis was not conducted.
Time Frame: During the infusion (single bolus dose of hylenex [1 hr], followed by subcutaneous fluid for 1 hour to 72 hours)
Population: Randomized Population. Only those participants who did not receive subcutaneous fluid administration by hylenex-facilitated infusion as rescue were to be analyzed.
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid: Non-rescued
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Mean Total Volume of Fluid Administered at All Infusion Sites, From the Start to the Cessation of Fluid Administration, for All Rescued Participants Achieving > 200 mL
Description: as for outcome 6
Time Frame: During the infusion (single bolus dose of hylenex [1 hr], followed by subcutaneous fluid for 1 hour to 72 hours)
Population: Randomized Participants. Only those participants randomized to receive intravenous isotonic fluid who received subcutaneous fluid administration by hylenex-facilitated infusion as rescue were analyzed.
Arm/Group | Intravenous Isotonic Fluid: SC Rescued
Number analyzed (Participants) | 0

8. Secondary Outcome: Mean Flow Rate, Delivered Per Unit Time, for All Randomized Participants
Description: The mean flow rate was averaged over any 60-minute period of time.
Time Frame: During the infusion (single bolus dose of hylenex [1 hr], followed by subcutaneous fluid for 1 hour to 72 hours)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: milliliters per hour
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid
Number analyzed (Participants) | 73 | 75
milliliters per hour
  Emergency department plus hospital stay | 183.8 (94.61) | 166.1 (142.52)
  Emergency department stay only | 186.4 (92.21) | 179.6 (141.19)
Statistical Analysis 1: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -30.1, 95% CI 2-sided [-69.5 to 9.4] — Treatment difference: subcutaneous minus intravenous; Emergency department plus hospital stay
Statistical Analysis 2: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -40.2, 95% CI 2-sided [-77.3 to -3.1] — Treatment difference: subcutaneous minus intravenous; Emergency department stay only

9. Secondary Outcome: Mean Flow Rate, Delivered Per Unit Time, for All Non-rescued Participants
Description: The mean flow rate was averaged over any 60-minute period of time. Participants randomized to receive intravenous isotonic fluid were permitted to receive subcutaneous fluid administration by hylenex-facilitated infusion as rescue.
Time Frame: During the infusion (single bolus dose of hylenex [1 hr], followed by subcutaneous fluid for 1 hour to 72 hours)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milliliters per hour
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid: Non-rescued
Number analyzed (Participants) | 73 | 59
milliliters per hour
  Emergency department plus hospital stay | 183.8 (94.61) | 211.1 (127.44)
  Emergency department stay only | 186.4 (92.21) | 228.3 (118.82)
Statistical Analysis 1: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid: Non-rescued; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -30.1, 95% CI 2-sided [-69.5 to 9.4] — Treatment difference: subcutaneous minus intravenous; Emergency department plus hospital stay
Statistical Analysis 2: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid: Non-rescued; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -40.2, 95% CI 2-sided [-77.3 to -3.1] — Treatment difference: subcutaneous minus intravenous; Emergency department stay only

10. Secondary Outcome: Mean Flow Rate, Delivered Per Unit Time, for All Rescued Participants
Description: as for outcome 9
Time Frame: During the infusion (single bolus dose of hylenex [1 hr], followed by subcutaneous fluid for 1 hour to 72 hours)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milliliters per hour
Arm/Group | Intravenous Isotonic Fluid: SC Rescued
Number analyzed (Participants) | 15
milliliters per hour
  Emergency department plus hospital stay | 139.1 (80.27)
  Emergency department stay only | 149.8 (79.53)

11. Secondary Outcome: Mean Flow Rate, Delivered by Volume Per Unit Body Weight Per Unit Time, for All Randomized Participants
Description: The mean flow rate was averaged over any 60-minute period of time.
Time Frame: During the infusion (single bolus dose of hylenex [1 hr], followed by subcutaneous fluid for 1 hour to 72 hours)
Population: ITT Population. Only those participants with evaluable data (known volume and known baseline body weight) were analyzed.
Measure: Mean (Standard Deviation); unit: milliliters per kilogram per hour
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid
Number analyzed (Participants) | 70 | 73
milliliters per kilogram per hour
  Emergency department plus hospital stay | 15.4 (5.62) | 12.3 (9.50)
  Emergency department stay only | 15.6 (5.33) | 13.3 (9.50)
Statistical Analysis 1: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.9, 95% CI 2-sided [0.3 to 5.5] — Treatment difference: subcutaneous minus intravenous; Emergency department plus hospital stay
Statistical Analysis 2: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.2, 95% CI 2-sided [-0.2 to 4.7] — Treatment difference: subcutaneous minus intravenous; Emergency department stay only

12. Secondary Outcome: Mean Flow Rate, Delivered by Volume Per Unit Body Weight Per Unit Time, for All Non-rescued Participants
Description: as for outcome 9
Time Frame: During the infusion (single bolus dose of hylenex [1 hr], followed by subcutaneous fluid for 1 hour to 72 hours)
Population: ITT Population. Only those participants who did not receive subcutaneous fluid administration by hylenex-facilitated infusion as rescue were analyzed. Only those participants with evaluable data (known volume and known baseline body weight) were analyzed.
Measure: Mean (Standard Deviation); unit: milliliters per kilogram per hour
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid: Non-rescued
Number analyzed (Participants) | 70 | 57
milliliters per kilogram per hour
  Emergency department plus hospital stay | 15.4 (5.62) | 15.7 (7.80)
  Emergency department stay only | 15.6 (5.33) | 17.1 (7.14)
Statistical Analysis 1: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid: Non-rescued; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-2.8 to 1.9] — Treatment difference: subcutaneous minus intravenous; Emergency department plus hospital stay
Statistical Analysis 2: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid: Non-rescued; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-3.4 to 0.8] — Treatment difference: subcutaneous minus intravenous; Emergency department stay only

13. Secondary Outcome: Mean Flow Rate, Delivered by Volume Per Unit Body Weight Per Unit Time, for All Rescued Participants
Description: as for outcome 9
Time Frame: During the infusion (single bolus dose of hylenex [1 hr], followed by subcutaneous fluid for 1 hour to 72 hours)
Population: ITT Population. Only those participants randomized to receive intravenous isotonic fluid who received subcutaneous fluid administration by hylenex-facilitated infusion as rescue were analyzed. Only those participants with evaluable data (known volume and known baseline body weight) were analyzed.
Measure: Mean (Standard Deviation); unit: milliliters per kilogram per hour
Arm/Group | Intravenous Isotonic Fluid: SC Rescued
Number analyzed (Participants) | 14
milliliters per kilogram per hour
  Emergency department plus hospital stay | 14.4 (6.47)
  Emergency department stay only | 15.4 (6.07)

14. Secondary Outcome: Number of Participants Achieving a Maximum Flow Rate of > 2 Milliliters Per Minute (mL/Min), as an Indication of Successful Hydration
Description: The maximum flow rate was averaged over any 60-minute period of time.
Time Frame: During the infusion (single bolus dose of hylenex [1 hr], followed by subcutaneous fluid for 1 hour to 72 hours)
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid
Number analyzed (Participants) | 73 | 75
Participants | 68 | 57

15. Secondary Outcome: Number of Participants Administered at Least 200 Milliliter (mL) Total Volume at a Single Infusion Site, From the Start to the Cessation of Fluid Administration
Description: The number of participants administered at least 20 mL total volume was assessed.
Time Frame: During the infusion (single bolus dose of hylenex [1 hr], followed by subcutaneous fluid for 1 hour to 72 hours)
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid
Number analyzed (Participants) | 73 | 75
Participants | 18 | 27

16. Secondary Outcome: Number of Participants With the Indicated Type of Adverse Events
Description: Adverse events (AEs) are defined as any untoward medical occurrence in a participant administered a product, which did not necessarily have a causal relationship with the treatment. Treatment-emergent adverse events (TEAEs) are defined as those events that occurred on or after the first injection device insertion attempt.
Time Frame: up to 7 days after hospital discharge
Population: Safety Population: all randomly assigned participants for whom the treatment was attempted (i.e., infusion device placement was initiated)
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid
Number analyzed (Participants) | 73 | 75
Participants
  At least 1 AE | 73 | 68
  At least 1 infusion site AE | 73 | 63
  at least 1 AE related to infusion fluid | 72 | 32
  At least 1 AE related to hylenex | 67 | 14

17. Secondary Outcome: Number of Participants With Normal Physical Examination Findings at Baseline That Shifted to Abnormal at the End of Fluid Administration
Description: Baseline was defined as the time prior to the single site fluid infusion. End of infusion was defined as the end of infusion of the single site fluid infusion for participants who had more than one fluid infusion. Not Rel Dehy = Abnormal, Not Related to Dehydration; Rel Dehy = Abnormal, Related to Dehydration. The investigator assessed findings as abnormal.
Time Frame: Baseline; after infusion (single bolus dose of hylenex [1 hr], followed by subcutaneous fluid for 1 hour to 72 hours)
Population: Safety Population. Only those participants for which fluid administration was initiated were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid: Non-rescued | Intravenous Isotonic Fluid: SC Rescued
Number analyzed (Participants) | 73 | 59 | 15
Participants
  Head, eyes, ears: Not Rel Dehy | 1 | 0 | 0
  Head, eyes, ears: Rel Dehy | 0 | 0 | 0
  Neck/upper airway: Not Rel Dehy | 0 | 0 | 0
  Neck/upper airway: Rel Dehy | 0 | 0 | 0
  Heart: Not Rel Dehy | 0 | 1 | 0
  Heart: Rel Dehy | 0 | 0 | 0
  Lungs: Not Rel Dehy | 0 | 0 | 0
  Lungs: Rel Dehy | 0 | 0 | 0
  Abdomen: Not Rel Dehy | 0 | 0 | 0
  Abdomen: Rel Dehy | 0 | 0 | 0
  Skin: Not Rel Dehy | 0 | 1 | 2
  Skin: Rel Dehy | 0 | 0 | 0
  Musculoskeletal: Not Rel Dehy | 0 | 0 | 0
  Musculoskeletal: Rel Dehy | 0 | 0 | 0
  Extremities: Not Rel Dehy | 0 | 0 | 0
  Extremities: Rel Dehy | 0 | 0 | 0
  Neurological: Not Rel Dehy | 1 | 0 | 0
  Neurological: Rel Dehy | 0 | 0 | 0
  Vascular/Circulatory: Not Rel Dehy | 0 | 0 | 0
  Vascular/Circulatory: Rel Dehy | 1 | 0 | 0
  Lymphatic: Not Rel Dehy | 0 | 0 | 0
  Lymphatic: Rel Dehy | 0 | 0 | 0
  Reproductive: Not Rel Dehy | 0 | 0 | 0
  Reproductive: Rel Dehy | 0 | 0 | 0
  Renal/Urinary: Not Rel Dehy | 0 | 0 | 0
  Renal/Urinary: Rel Dehy | 1 | 0 | 0
  Endocrine/Metabolism and Nutrition: Not Rel Dehy | 0 | 0 | 0
  Endocrine/Metabolism and Nutrition: Rel Dehy | 0 | 0 | 0
  Other: Not Rel Dehy: number analyzed (Participants) | 8 | 8 | 4
  Other: Not Rel Dehy | 0 | 0 | 0
  Other: Rel Dehy: number analyzed (Participants) | 8 | 8 | 4
  Other: Rel Dehy | 0 | 0 | 0

18. Secondary Outcome: Mean Change From Baseline in Heart Rate
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Baseline was defined as the time prior to the single site fluid infusion. End of infusion was defined as the end of infusion of the single site fluid infusion for participants who had more than one fluid infusion.
Time Frame: Baseline; after infusion (single bolus dose of hylenex [1 hr], followed by subcutaneous fluid for 1 hour to 72 hours)
Population: Safety Population. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid: Non-rescued | Intravenous Isotonic Fluid: SC Rescued
Number analyzed (Participants) | 68 | 53 | 14
beats per minute | -6.9 (17.38) | -4.8 (18.64) | -11.3 (24.68)

19. Secondary Outcome: Mean Change From Baseline in Respiratory Rate
Description: as for outcome 18
Time Frame: Baseline; after infusion (single bolus dose of hylenex [1 hr], followed by subcutaneous fluid for 1 hour to 72 hours)
Population: Safety Population. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid: Non-rescued | Intravenous Isotonic Fluid: SC Rescued
Number analyzed (Participants) | 68 | 52 | 14
breaths per minute | -4.8 (9.76) | -1.3 (7.96) | -2.6 (13.36)

20. Secondary Outcome: Mean Change From Baseline in Systolic Blood Pressure and Diastolic Blood Pressure
Description: as for outcome 18
Time Frame: Baseline; after infusion (single bolus dose of hylenex [1 hr], followed by subcutaneous fluid for 1 hour to 72 hours)
Population: Safety Population. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid: Non-rescued | Intravenous Isotonic Fluid: SC Rescued
Number analyzed (Participants) | 61 | 49 | 14
millimeters of mercury (mmHg)
  Systolic blood pressure | 3.2 (16.15) | 1.1 (15.49) | -4.0 (24.17)
  Diastolic blood pressure | -0.2 (12.43) | 0.7 (12.45) | -2.9 (23.07)

21. Secondary Outcome: Mean Change From Baseline in the Face, Legs, Activity, Cry, Consolability (FLACC) Pain Scale Score
Description: The infusion site was assessed for pain at two time points: after placement of the infusion device but before fluid infusion and at the end of infusion. Pain was recorded using the FLACC pain scale for children less than 3 years of age. Scores on the scale ranged from 0 (no hurt) to 10 (hurt worst).
Time Frame: Before infusion (Baseline); after infusion (single bolus dose of hylenex [1 hr], followed by subcutaneous fluid for 1 hour to 72 hours)
Population: Safety Population. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid: Non-rescued | Intravenous Isotonic Fluid: SC Rescued
Number analyzed (Participants) | 59 | 39 | 15
score on a scale | -4.4 (3.45) | -5.2 (2.94) | -3.8 (2.11)

22. Secondary Outcome: Number of Participants With the Indicated Type of Fluid Administered
Description: Data are reported for the initial fluid administered.
Time Frame: During the infusion (single bolus dose of hylenex [1 hr], followed by subcutaneous fluid for 1 hour to 72 hours)
Population: ITT Population. Only those participants for which fluid administration was initiated were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid: Non-rescued | Intravenous Isotonic Fluid: SC Rescued
Number analyzed (Participants) | 73 | 59 | 15
Participants
  Lactated Ringers | 28 | 9 | 6
  Normal saline (NS) | 44 | 49 | 9
  D5 1/2 NS without potassium chloride (KCL) | 0 | 1 | 0
  D5 1/2 NS with KCL | 0 | 0 | 0
  Other | 1 | 0 | 0

23. Secondary Outcome: Infusion Duration During the Initial Infusion
Description: Infusion duration was assessed as a measure of the time required to complete the initial infusion of 20 mL/kg.
Time Frame: first hour of infusion
Population: ITT Population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid
Number analyzed (Participants) | 73 | 75
hours | 1.0 (0.13) | 0.8 (0.42)
Statistical Analysis 1: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid; Test type: Superiority; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [0.1 to 0.3] — Treatment difference = SC minus IV

24. Secondary Outcome: Change From Baseline in Hydration Status According to the Gorelick Assessment at the End of Fluid Infusion
Description: Hydration status was assessed clinically using the Gorelick 10-item scale: general condition, quality of radial pulse, quality of respiration, skin elasticity, eyes, tears, mucous membranes, urine output, heart rate, and capillary refill time at the fingertip. Scores ranged from 0 (less severe impairment) to 10 (more severe impairment). Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; during the infusion (single bolus dose of hylenex [1 hr], followed by subcutaneous fluid for 1 hour to 72 hours)
Population: ITT Population. Only those participants contributing data at the indicated time point were assessed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid
Number analyzed (Participants) | 73 | 73
score on a scale | -2.6 (1.26) | -2.2 (1.64)
Statistical Analysis 1: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid; Test type: Superiority; p = 0.0658, ANOVA; From Analysis of Variance (ANOVA) model with center and treatment as factors; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.9 to 0.0] — Treatment difference = SC minus IV

25. Secondary Outcome: Percent Change From Baseline in Body Weight
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] / Baseline value) * 100.
Time Frame: as for outcome 24
Population: ITT Population. Only those participants contributing data at the indicated time point were assessed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid
Number analyzed (Participants) | 68 | 67
percent change | 2.9 (2.52) | 3.8 (15.17)
Statistical Analysis 1: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid; Test type: Superiority; p = 0.6208, ANOVA; From ANOVA model with center and treatment as factors; Mean Difference (Net) = -1.0, 95% CI 2-sided [-4.8 to 2.9] — Treatment difference = SC minus IV

26. Secondary Outcome: Number of Participants With the Indicated Type of Rescue Route Therapy Administered
Description: Participants for whom parenteral access by the randomized route of administration could not be achieved after a reasonable number of attempts and for whom the investigator had deemed the access by that route a failure were expected to receive fluid administration by other means, designated as "rescue route" for the purpose of this study. This rescue route may have included venous cut-down, central venous line, interosseous access, etc., and for those participants initially randomly assigned to IV fluid administration, SC fluid administration by hylenex-facilitated infusion.
Time Frame: During the infusion (single bolus dose of hylenex [1 hr], followed by subcutaneous fluid for 1 hour to 72 hours)
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid
Number analyzed (Participants) | 73 | 75
Participants
  hylenex-facilitated SC | 0 | 15
  Other type of rescue | 0 | 0

27. Secondary Outcome: Number of Participants Classified With the Indicated Healthcare Provider Responses to the Questions Comprising the Healthcare Provider Global Satisfaction Questionnaire
Description: A global assessment of overall satisfaction with the rehydration therapy by healthcare provider was performed at the end of SC or IV fluid rehydration utilizing a simple questionnaire. There were separate questionnaires for the two types of rehydration (SC and IV). Question 1: Was the participant successfully hydrated using the randomized route of administration?; Question 2: Overall, was the procedure of fluid infusion easy to perform?; Question 3: Were there any unacceptable side effects from the therapy?; Question 4: Would you consider using this hydration therapy for this indication in the future?
Time Frame: During the infusion (single bolus dose of hylenex [1 hr], followed by subcutaneous fluid for 1 hour to 72 hours)
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid
Number analyzed (Participants) | 73 | 75
Participants
  Question 1: Yes | 68 | 57
  Question 1: No | 4 | 13
  Question 1: Missing | 1 | 5
  Question 2: Yes | 69 | 49
  Question 2: No | 4 | 21
  Question 2: Missing | 0 | 5
  Question 3: Yes | 3 | 4
  Question 3: No | 70 | 66
  Question 3: Missing | 0 | 5
  Question 4: Yes | 71 | 64
  Question 4: No | 2 | 6
  Question 4: Missing | 0 | 5
Statistical Analysis 1: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid; Test type: Superiority; p = 0.0685, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel (CMH) test controlling for center; Question 1
Statistical Analysis 2: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid; Test type: Superiority; p = 0.0004, Cochran-Mantel-Haenszel — CMH test controlling for center; Question 2
Statistical Analysis 3: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid; Test type: Superiority; p = 0.6861, Cochran-Mantel-Haenszel — CMH test controlling for center; Question 3
Statistical Analysis 4: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid; Test type: Superiority; p = 0.2323, Cochran-Mantel-Haenszel — CMH test controlling for center; Question 4

28. Secondary Outcome: Number of Participants Classified With the Indicated Healthcare Provider Responses to the Question: How Does This Therapy Compare to Your Experience With IV (for SC Group) / SC (for IV Group) Therapy?
Description: A global assessment of overall satisfaction with the rehydration therapy by healthcare provider was performed at the end of SC or IV fluid rehydration utilizing a simple questionnaire. There were separate questionnaires for the two types of rehydration (SC and IV).
Time Frame: During the infusion (single bolus dose of hylenex [1 hr], followed by subcutaneous fluid for 1 hour to 72 hours)
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid
Number analyzed (Participants) | 73 | 75
Participants
  Effectiveness: Less Effective | 3 | 1
  Effectiveness: Same Effectiveness | 58 | 41
  Effectiveness: More Effective | 11 | 0
  Effectiveness: Missing | 1 | 0
  Degree of Difficulty: Less Difficult | 57 | 2
  Degree of Difficulty: Same Difficulty | 11 | 12
  Degree of Difficulty: More Difficult | 3 | 28
  Degree of Difficulty: Missing | 2 | 0
  Not applicable: no prior experience with alternate | 0 | 33
Statistical Analysis 1: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid; Test type: Superiority; p = 0.0033, Cochran-Mantel-Haenszel — CMH test controlling for center; Effectiveness
Statistical Analysis 2: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — CMH test controlling for center; Degree of difficulty

29. Secondary Outcome: Number of Participants Classified With the Indicated Parent/Guardian Responses to the Questions Comprising the Parent / Guardian Global Satisfaction Questionnaire
Description: A global assessment of overall satisfaction with the rehydration therapy by healthcare provider was performed at the end of SC or IV fluid rehydration utilizing a simple questionnaire. There were separate questionnaires for the two types of rehydration (SC and IV). Question 1: Do you believe the method of therapy was successful in your child's rehydration?; Question 2: Have you or your child ever previously had IV fluids (for SC Group) / SC fluids (for IV Group)?; Question 3: If the response to Question 2 was "yes," how does this compare to prior experience with IV (for SC Group) / SC (for IV Group)?; Question 4: Should your child(ren) need rehydration treatment in the future, would you opt for this procedure?; Question 5: Should you need rehydration treatment in the future, would you opt for this procedure?; Question 6: What is your global satisfaction with the study procedure?
Time Frame: During the infusion (single bolus dose of hylenex [1 hr], followed by subcutaneous fluid for 1 hour to 72 hours)
Population: ITT Population. Only participants with a response of "Yes" to Question 2 contributed responses for Question 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid
Number analyzed (Participants) | 73 | 75
Participants
  Question 1, yes | 70 | 59
  Question 1, no | 3 | 8
  Question 1, missing | 0 | 8
  Question 2, yes | 47 | 2
  Question 2, no | 26 | 63
  Question 2, not done | 0 | 2
  Question 2, missing | 0 | 8
  Question 3, worse: number analyzed (Participants) | 73 | 2
  Question 3, worse | 2 | 0
  Question 3, same: number analyzed (Participants) | 73 | 2
  Question 3, same | 9 | 2
  Question 3, better: number analyzed (Participants) | 73 | 2
  Question 3, better | 35 | 0
  Question 3, missing: number analyzed (Participants) | 73 | 2
  Question 3, missing | 1 | 0
  Question 4, yes | 65 | 56
  Question 4, no | 4 | 11
  Question 4, not done | 2 | 0
  Question 4, unknown | 1 | 0
  Question 4, missing | 1 | 8
  Question 5, yes | 68 | 55
  Question 5, no | 4 | 12
  Question 5, not done | 1 | 0
  Question 5, missing | 0 | 8
  Question 6, very unsatisfied | 3 | 8
  Question 6, unsatisfied | 1 | 4
  Question 6, satisfied | 26 | 31
  Question 6, very satisfied | 43 | 24
  Question 6, missing | 0 | 8
Statistical Analysis 1: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid; Test type: Superiority; p = 0.2012, Cochran-Mantel-Haenszel — CMH test controlling for Center; Question 1
Statistical Analysis 2: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — CMH test controlling for center; Question 2
Statistical Analysis 3: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid; Test type: Superiority; p = 0.1302, Cochran-Mantel-Haenszel — CMH test controlling for center; Question 4
Statistical Analysis 4: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid; Test type: Superiority; p = 0.0852, Cochran-Mantel-Haenszel — CMH test controlling for center; Question 5
Statistical Analysis 5: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid; Test type: Superiority; p = 0.0275, Cochran-Mantel-Haenszel — CMH test controlling for center; Question 6

30. Secondary Outcome: Number of Participants With the Indicated Number of Different Anatomical Administration Sites Needed After the Start of Fluid Administration
Description: In the event that the degree of local infusion site swelling became unacceptable for any reason (e.g., a 30% or greater increase from the baseline circumference of the infused thigh or in the clinical judgment of the investigator), the infusion rate was decreased or the infusion site was changed.
Time Frame: During the infusion (single bolus dose of hylenex [1 hr], followed by subcutaneous fluid for 1 hour to 72 hours)
Population: ITT Population. Only those participants for which fluid administration was initiated were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid: Non-rescued | Intravenous Isotonic Fluid: SC Rescued
Number analyzed (Participants) | 73 | 59 | 15
Participants
  1 administration site | 72 | 59 | 15
  2 administration sites | 1 | 0 | 0

31. Secondary Outcome: Number of Participants Experiencing Reductions in Flow Rate
Description: as for outcome 30
Time Frame: During the infusion (single bolus dose of hylenex [1 hr], followed by subcutaneous fluid for 1 hour to 72 hours)
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid
Number analyzed (Participants) | 73 | 75
Participants | 43 | 39

32. Secondary Outcome: Number of Participants Who Received Needle Placement by People With the Indicated Level of Staff Training
Description: Data were collected for the level of staff training for the person who performed the needle placement.
Time Frame: average of approximately 3 minutes
Population: ITT Population. Only those participants for which fluid administration was initiated were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid: Non-rescued | Intravenous Isotonic Fluid: SC Rescued
Number analyzed (Participants) | 73 | 59 | 15
Participants
  Physician | 28 | 4 | 1
  Registered nurse | 35 | 48 | 10
  Physician assistant | 2 | 2 | 1
  Nurse practitioner | 6 | 0 | 0
  Licensed vocational nurse | 0 | 0 | 2
  Other | 2 | 5 | 1

33. Secondary Outcome: Number of Participants for Which the Indicated Number of Additional Personnel Was Involved in Needle Placement
Description: Data were collected for the number of additional personnel involved in needle placement.
Time Frame: average of approximately 3 minutes
Population: ITT Population. Only those participants for which fluid administration was initiated were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid: Non-rescued | Intravenous Isotonic Fluid: SC Rescued
Number analyzed (Participants) | 73 | 59 | 15
Participants
  0 | 20 | 1 | 1
  1 | 36 | 34 | 5
  2 | 14 | 20 | 7
  3 | 3 | 3 | 2
  4 | 0 | 1 | 0

34. Secondary Outcome: Time From the Start of Infusion to the Time of Emergency Department (ED) Discharge
Description: Data are reported from the start of infusion to the time of ED discharge.
Time Frame: up to approximately 26 hours
Population: ITT Population. Only those participants for which fluid administration was initiated were analyzed. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid: Non-rescued | Intravenous Isotonic Fluid: SC Rescued
Number analyzed (Participants) | 72 | 59 | 15
hours | 4.0 (4.26) | 3.1 (1.92) | 4.7 (4.64)

35. Secondary Outcome: Time From Randomization to the First Drop of Fluid Infusion
Description: Data are reported for the time from randomization to the start of fluid infusion for all randomized participants.
Time Frame: up to approximately 110 and 220 minutes for the SC and IV arms, respectively
Population: ITT Population. Only those participants for which fluid administration was initiated were analyzed.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid
Number analyzed (Participants) | 73 | 74
minutes | 37 [31 to 41] | 42.5 [37 to 52]
Statistical Analysis 1: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid; Test type: Superiority; p = 0.0247, Wilcoxon (Mann-Whitney)

36. Secondary Outcome: Number of Participants With the Indicated Number of Needle Stick Attempts Needed to Initiate Fluid Administration
Description: Data are reported for the number of needle stick attempts needed to initiate fluid administration.
Time Frame: average of approximately 3 minutes
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid
Number analyzed (Participants) | 73 | 75
Participants
  1 | 69 | 54
  2 | 4 | 13
  3 | 0 | 7
  >3 | 0 | 1
Statistical Analysis 1: Comparison: Subcutaneous Hylenex vs Intravenous Isotonic Fluid; Test type: Superiority; p = 0.0007, Cochran-Mantel-Haenszel — CMH test controlling for center

37. Secondary Outcome: Number of Participants for Which the Indicated Type of Infusion Device Was Used
Description: Data are reported for the type of infusion device used.
Time Frame: average of approximately 3 minutes
Population: ITT Population. Only those participants for which fluid administration was initiated were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid: Non-rescued | Intravenous Isotonic Fluid: SC Rescued
Number analyzed (Participants) | 73 | 59 | 15
Participants
  Angiocatheter | 63 | 57 | 15
  Butterfly needle | 10 | 1 | 0
  Other | 0 | 1 | 0

38. Secondary Outcome: Number of Participants for Which the Indicated Gauge for Infusion Device Was Used
Description: Data are reported for the gauge of infusion device used.
Time Frame: average of approximately 3 minutes
Population: ITT Population. Only those participants for which fluid administration was initiated were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid: Non-rescued | Intravenous Isotonic Fluid: SC Rescued
Number analyzed (Participants) | 73 | 59 | 15
Participants
  20 | 2 | 0 | 0
  22 | 28 | 22 | 5
  23 | 4 | 1 | 0
  24 | 31 | 33 | 10
  25 | 8 | 2 | 0
  26 | 0 | 1 | 0

39. Secondary Outcome: Number of Participants Discharged From the ED to Home or the Hospital
Description: Participants were discharged from the ED to home or the hospital to continue hydration therapy.
Time Frame: up to approximately 26 hours
Population: ITT Population. Only those participants for which fluid administration was initiated were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid
Number analyzed (Participants) | 73 | 74
Participants
  Home | 60 | 64
  Hospital | 13 | 10

40. Secondary Outcome: Number of Participants With the Indicated Reason for Rehospitalization Within 48 and 72 Hours After Discharge
Description: Participants were discharged from the ED to home or the hospital to continue hydration therapy.
Time Frame: from randomization up to approximately 98 hours
Population: ITT Population. Only those participants who were re-hospitalized or had an Emergency Department visit after initial discharge to home were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid
Number analyzed (Participants) | 9 | 10
Participants
  Retreatment for dehydration | 2 | 2
  Other | 7 | 8

ADVERSE EVENTS:
Description: Adverse event data are reported in members of the Safety Population, comprised of all randomly assigned participants for whom the treatment was attempted (i.e., infusion device placement was initiated)
Arm/Group | Subcutaneous Hylenex | Intravenous Isotonic Fluid
All-Cause Mortality (participants affected / at risk) | 1/73 | 0/75
Serious Adverse Events (participants affected / at risk) | 3/73 | 4/75
Other Adverse Events (participants affected / at risk) | 73/73 | 62/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subcutaneous Hylenex (N=73) | Intravenous Isotonic Fluid (N=75)
Pyrexia (General disorders) | 0 | 1
Ongoing dehydration (Metabolism and nutrition disorders) | 0 | 1
Rotavirus infection (Infections and infestations) | 0 | 1
Kawasaki disease (Vascular disorders) | 0 | 1
Viral gastroenteritis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Cardio-respiratory Arrest (Cardiac disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Subcutaneous Hylenex (N=73) | Intravenous Isotonic Fluid (N=75)
Infusion site erythema (General disorders) | 54 | 19
Infusion site haematoma (General disorders) | 0 | 3
Infusion site oedema (General disorders) | 5 | 1
Infusion site pain (General disorders) | 57 | 59
Infusion site swelling (General disorders) | 59 | 16
Pyrexia (General disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information obtained as a result of this study or during the conduct of this study will be regarded as confidential. The Investigator agrees to use the information for the purpose of carrying out this study and for no other purpose, unless written permission from the sponsor (Halozyme) is obtained.